CLINICAL TRIAL: NCT02123264
Title: Randomized Clinical Trial on the Prevention of Radiographic Progression With Zoledronic Acid in Patients With Early Rheumatoid Arthritis and Low Disease Activity
Brief Title: Zoledronic Acid in Rheumatoid Arthritis
Acronym: AZAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Carmen Gómez-Vaquero (Other)
Responsible Party: Sponsor-Investigator, Carmen Gómez-Vaquero, MD PhD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CGV222
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid (Active Comparator): Zoledronic acid: 5 mg/year x 2 years
  Interventions: Drug: Zoledronic acid
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid: 5 mg/year x 2 years
  Other Names: Aclasta
  Arms: Zoledronic acid

SUMMARY:
The progression of structural joint damage is the leading cause of disability and socioeconomic costs associated with rheumatoid arthritis (RA). Remission and low clinical activity not always imply absence of progression of structural damage. The main objective of this study is to evaluate the progression of radiological damage in early RA patients currently treated with disease modifying anti-rheumatic drugs (DMARDs) and low disease activity to which treatment with zoledronic acid is added.

The investigators propose a randomized clinical trial in 94 patients with RA of less than 2 years of evolution that, being treated with DMARDs, present criteria of low disease activity (DAS28 < 3.2).

Patients will be randomized into two branches: zoledronic acid and no treatment. The primary study endpoint is the progression of radiological damage assessed in a blinded way by the difference in the Sharp-van der Heijde index (SHI) in radiographs of hands and feet after two years; the secondary variables: radiographic progression after one year, serum bone biomarkers (OPG, RANKL, DKK-1 and sclerostin) and adverse effects. In a subgroup of patients, the investigators shall evaluate the change in the size of hand erosions by multislice computed tomography and the evolution of periarticular osteoporosis and systemic bone mass by dual X-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 18 years
2. Patients with RA of less than 2 years of evolution
3. DMARD therapy (methotrexate alone or methotrexate, leflunomide or methotrexate within COBRA strategy) on stable dose for at least 6 weeks prior to study entry
4. Patients not treated with glucocorticoids or under stable dose of prednisone up to 5 mg / day or equivalent dose of another glucocorticoid
5. Low disease activity (DAS28 <3.2)
6. In case of premenopausal women, commitment to make contraceptive treatment up to 3 years after the last dose of zoledronic acid
7. Signed informed consent

Exclusion Criteria:

1. Previous or current treatment with biological drugs used for the treatment of RA (infliximab, adalimumab, etanercept, certolizumab, golimumab, rituximab, abatacept, tocilizumab)
2. Pretreatment with:

   1. Bisphosphonates in the 5 years prior to the onset of RA
   2. Calcitonin, raloxifene, bazedoxifene, strontium ranelate, teriparatide and denosumab in the year before the onset of RA
3. Contraindication to treatment with zoledronic acid:

   1. Hypersensitivity to bisphosphonates
   2. Hypocalcemia
   3. Glomerular filtration rate <35 mL / min
   4. Pregnant (negative pregnancy test) and lactating women
   5. Poor oral hygiene
   6. Pending invasive dental procedure
4. Serum levels of calcidiol lower than 25 nmol/L (10 ng/mL).
5. Simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Sharp van der Heijde index | Two years
  To assess the progression of radiographic damage in patients with early RA in current treatment with DMARDs and low disease activity to which treatment with zoledronic acid is added, compared to a no treatment control population, after two years.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez-Vaquero, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge; Silvia Pérez-Pujol, PhD, Study Director — UCICEC-Hospital Universitari de Bellvitge
Locations (11):
- Spain (11):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Sant Joan Despí Moisés Broggi, Sant Joan Despí, Barcelona
  - Hospital Residència Sant Camil, Sant Pere de Ribes, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bilbao
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen Macarena, Seville